CLINICAL TRIAL: NCT03940768
Title: The Use of Lactobacillus Plantarum 299v in Treatment of Cancer Patients Who Received Home Enteral Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Karolina Kaźmierczak-Siedlecka, Karolina Kaźmierczak-Siedlecka (nutritionist, PhD student - Department of Surgical Oncology), Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUGdansk1
Record Dates: First submitted 2019-01-31; First posted 2019-05-07 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: cancer; home enteral nutrition; probiotic; Lactobacillus plantarum 299v
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum 299v receivers (Experimental): Sanprobi IBS (Lactobacillus plantarum 299v) 2 capsules per day for 4 weeks.
  Interventions: Dietary Supplement: Lactobacillus plantarum 299v; Dietary Supplement: Placebo
- Placebo receivers (Placebo Comparator): Sanprobi IBS placebo 2 capsules per day for 4 weeks.
  Interventions: Dietary Supplement: Lactobacillus plantarum 299v; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum 299v — Administration of Lactobacillus plantarum 299v in cancer patients who receive home enteral nutrition.
Dietary Supplement: Placebo — Administration of placebo in cancer patients who receive home enteral nutrition.

SUMMARY:
The aim of the study is to assess the impact of Lactobacillus plantarum 299v on nutritional status, tolerance of enteral diet and the quality of life. Administration of this probiotic may potentially improve nutritional status and tolerance of enteral diet. It also may provide positive effect on quality of life.

DETAILED DESCRIPTION:
Study group consists of patients with cancer who are qualified for home enteral nutrition in Nutritional Counselling Center Copernicus in Gdansk. The control group will receive home enteral nutrition and placebo. The experimental group will receive home enteral nutrition and Lactobacillus plantarum 299v. The study is prospective and double-blind. The parameters for evaluation of nutritional status are: BMI, body mass analysis, level of total protein and albumin in blood serum, total lymphocyte count, NRS 2002 method. Assessment of the quality of life and tolerance of enteral diet will be done by questionaires.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 yr.,
* the presence of cancer, artificial access to the alimentary tract (naso-gastric tube, gastrostomy, percutaneous endoscopic gastrostomy, jejunostomy, microjejunostomy),
* qualification for home enteral nutrition,
* written consent to take part in the study

Exclusion Criteria:

* age <18 yr.,
* patients requiring home parenteral nutrition,
* patients who are not being able to attend the visit in the study centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Changes of fat mass | at baseline and after 4th week
  fat mass in percent (%)
Changes of muscle mass | at baseline and after 4th week
  muscle mass in kilograms (kg)
Changes of total body water | at baseline and after 4th week
  total body water in percent (%)
Changes of body mass index | at baseline and after 4th week
  body mass index in kg/m^2
Changes of the albumin concentration | at baseline and after 4th week
  albumin concentration g/L
Changes of total protein concentration | at baseline and after 4th week
  total protein concentration g/L
Changes of total lymphocyte count | at baseline and after 4th week
  number of total lymphocyte count/mm^3

SECONDARY OUTCOMES:
Change of enteral nutrition tolerance | it will be filled every day by patients per 4 weeks treatment period
  The enteral nutrition tolerance will be assessed with authors own questionnaire referring to number of stools, frequency of vomiting and flatulence.
Change of patients' quality of life ( BREF - WHOQOL - Bref The World Health Organization Quality of Life) | at baseline and after 4th week
  Questionare containing questions divided in 4 domains (regarding environment, psychological, somatic, social factors). Each question gets points in scale 1-5, where 1 being the worst score. Within each domain poins are summed up.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutritional Counselling Centre Copernicus in Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kazmierczak-Siedlecka K, Folwarski M, Skonieczna-Zydecka K, Ruszkowski J, Makarewicz W. The use of Lactobacillus plantarum 299v (DSM 9843) in cancer patients receiving home enteral nutrition - study protocol for a randomized, double-blind, and placebo-controlled trial. Nutr J. 2020 Sep 11;19(1):98. doi: 10.1186/s12937-020-00598-w. PMID 32917221